CLINICAL TRIAL: NCT04446936
Title: A Retrospective Study Comparing Failure and Complications Rates Between Propeller Flap and Random Flap for Pressure Ulcer
Brief Title: Comparing Different Surgical Techniques for Coverage of Pressure Ulcer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0366
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Pressure Ulcer
Keywords: Ulcer; Flap; Random; Propeller; Paraplegic; Surgery
MeSH Terms: conditions — Pressure Ulcer; Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Propeller flaps: Patients who undergone propeller flap surgery
  Interventions: Procedure: Flap covering for pressure ulcer
- Random flaps: Patients who undergone random flap surgery
  Interventions: Procedure: Flap covering for pressure ulcer

INTERVENTIONS:
Procedure: Flap covering for pressure ulcer — Flap covering for pressure ulcer

SUMMARY:
The Plastic, Reconstructive and Aesthetic Surgery department of Montpellier was born out of the Wound and Healing department, the first unit of this type to be created in Europe. The investigators quickly became the national leader in the management of pressure ulcers, especially in people with spinal cord injuries.

Our expertise has evolved over time as well as our surgical techniques for covering ulcers, gradually over time the investigators have gone from " random " flaps to " propeller " flaps, more reliable in terms of vascularization and more logical in terms of force distribution and skin tension.

The investigators found subjectively that the rate of complications was lower for the helical flaps. The investigators therefore seek to confirm this trend through a retrospective study on patients operated on in the department between January 1, 2015 and December 31, 2019.

ELIGIBILITY:
Inclusion criteria:

* Major Patient
* Patient with trochanteric, ischiatic or sacral pressure ulcer
* Patient who undergone flap surgery for pressure ulcer between January 1st, 2015 and December 31st, 2019

Exclusion criteria:

* Other loss of substance than pressure ulcer
* Combined covering with a random flap and a propeller flap
* Surgical revision of a flap without a new flap

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sacral, trochanteric or ischiatic pressure ulcer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2021-01-20 (Estimated)

PRIMARY OUTCOMES:
Failure rate | 1 day
  Comparing failure rates between the two surgical techniques

SECONDARY OUTCOMES:
Complications rate | 1 day
  Comparing complications rate between the two surgical techniques

CONTACTS AND LOCATIONS:
Overall Officials: Farid BEKARA, MD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC